CLINICAL TRIAL: NCT01369992
Title: Molecular Profiling of Metastatic Cancer in Pleural Effusion and Ascites
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Tze-Sian Chan, Department of Gastroenterology
Other Study IDs: 99048
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Metastatic Cancer
Keywords: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Cancers are among the most frequent leading causes of death in Taiwan, and many of them show their respective unique epidemiological and pathophysiological features in Taiwanese population. One of the distinguishing features of cancers includes their potential to metastasize outside the primary tumor. Pleural cavity and peritoneum are two of the most frequent sites of metastases when serosal surfaces are involved. The prognoses of such patients are extremely poor with a median survival of months. The understandings of cancer biology of tumor metastasis demand more in-depth studies at the molecular and cell levels. Studies based on cell culture are excellent approaches for this purpose as the cell culture provides a relevant and renewable model for studying the pathological and molecular changes underlying human malignant tumors.

DETAILED DESCRIPTION:
Due to their easy accessibility, pleural effusions and ascites are two important clinical sources of metastatic cancer cells, which upon isolation, permit comparative studies between the biology nature of primary tumor and metastatic ones. In this study, we will try to isolate cancer cells from human malignant effusions, said to be pleural effusions and/or ascites. We will establish phenotypic alterations along the progression of malignant tumors with serosal metastasis, with special emphasis on expression of some proteases, laminin receptors and transcription factors involved in the process of invasion and metastasis. We would also perform clinical correlations, including tumor type, staging, status of lymph node metastasis and histopathological differentiation and grading, etc.

ELIGIBILITY:
Inclusion Criteria:

* cancer patients
* pleural effusion or peritoneal effusion

Exclusion Criteria:

* infected and fever patients
* anticoagulant treatment patients
* patients don't attend this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-05; Study Completion 2013-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tze-Sian Chan, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan